CLINICAL TRIAL: NCT01269944
Title: Effects of Osteotomies Around the Knee on Cartilage Glycosaminoglycan Content Using dGEMRIC Non-invasive Imaging, a Pilot Study
Brief Title: Effects of Osteotomies Around the Knee on Cartilage Glycosaminoglycan Content Using dGEMRIC Non-invasive Imaging
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, D.B.F. Saris, Prof. dr., UMC Utrecht
Other Study IDs: dGEMRIC HTO
Record Dates: First submitted 2010-12-29; First posted 2011-01-04 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Medial Compartment Osteoarthritis of the Knee
Keywords: osteoarthritis; knee; high wedge tibial osteotomy; dGEMRIC
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Medial compartment knee osteoarthritis: Patients with medial compartment osteoarthritis of the knee, as proven by x-rays and clinical examination

SUMMARY:
Medial compartment osteoarthritis of the knee is commonly treated by a surgical intervention called 'high tibial osteotomy' (VTO). Although it has repeatedly been shown that pain improves following this procedure, it is unknown how cartilage quality is affected by the procedure. In this study, a recently developed MRI technique is used to evaluate changes in cartilage quality before and after the surgery. Changes in MRI signals are correlated to subjective improvements (score lists). 10 patients participate in this study. Approval has been granted by the Medical Ethical Committee of the University Medical Center Utrecht. All participants are required to give informed consent before participation.

DETAILED DESCRIPTION:
Rationale: Medial compartment osteoarthritis (OA) of the knee is an invalidating disorder and leads to pain, decreased range of motion and inactivity. Two procedures aiming at maintaining original cartilage are the high tibial osteotomy (HTO) and the femur osteotomy. However, effects of this procedure on cartilage quality are not known.

Recently, a new technique has been developed which enables analysing changes in cartilage composition in vivo: the dGEMRIC. The dGEMRIC-technique is based on binding of negatively charged contrast agent Gadolinium (Gd(DPTA)2) to the glycosaminoglycans in the knee cartilage. The T1-signal reflects the gadolinium uptake by the proteoglycans of the knee and thus provides us with an indicative parameter of the cartilage quality. Visualising changes in cartilage composition enables better pre-operative patient selection as well as optimal timing of the operative procedure.

Objective: Primary objective: Evaluate changes in cartilage glycosaminoglycan content using dGEMRIC, in patients with osteoarthritis of the knee undergoing axial correction (HTO, femur osteotomy). Secondary objective: Correlate quantitative MRI data to subjective symptom scores (KOOS, WOMAC, VAS, Knee Society Score)

Study design: This study is a prospective observational study.

Study population: Ten patients will be included satisfying the following inclusion criteria:

* Both males and females older than 18 years
* Indication as set by treating physician for operative procedure around the knee: HTO (high tibial osteotomy), femoral osteotomy

Main study parameters/endpoints: In addition to their regular treatment, patients will receive an MRI scan with dGEMRIC settings before and 9 months after the surgical procedure, after removal of orthopaedic hardware. They will further receive questionnaires (VAS, WOMAC, KOOS, Knee Society Scale) before the surgical procedure and at 6,12, and 24 months after the surgical procedure.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In addition to their regular treatment, patients participating in this study will undergo two MRI scans of their knee. Performing of these scans will take about 4 hours. Further, orthopaedic hardware will be removed in daycare before the second MRI (burden: 1 day). Patients are asked to fill out questionnaires before- and after their surgical treatment. Filling out these questionnaires will take around 20 minutes per time moment (4 in total). Risks associated with the MRI scan are the very infrequently occurring allergic reactions to the contrast agent, which is used to depict the cartilage. Risks associated with removal of orthopaedic hardware at 9 months and not different than removal of hardware at a later stage: infection, bleeding, allergic reaction, dental damage or paresthesias.

ELIGIBILITY:
Inclusion Criteria:

Ten patients will be included satisfying the following inclusion criteria:

* Both males and females
* Patients >18 years old
* Indication as set by treating physician for operative procedure around the knee: HTO (high tibial osteotomy), femoral osteotomy
* Patient informed consent signed Note: Patients with previous surgery, history of intra-articular medication, meniscectomy or ACL lesions can be included in this study.

Exclusion Criteria:

* The following patients are excluded from participating in this study:
* Known anaphylactic reactions to Gadolinium or related substances
* Kidney diseases with a creatinin excretion of < 20 ml/min
* Risk groups for MRI scanning due to magnetic field or contrast agent (9, 10): Metal in body: Pacemaker / AICD / ICD (coronary defibrillator), Nervus vagus (X) stimulator, Artificial heart valve (depending on type), Metal clips on cerebral arteries or veins, Metal particles in eye, Port-a-cath, Metal stents, Hydrocephalic pump / insuline pump, Metal implants; f/e screws, prostheses, piercings.
* Claustrofibia
* First three months of pregnancy (not sufficient information available about effects of contrast agent on foetal development in this stage). Patients will be asked if they may be pregnant (< 3 months of pregnancy): if uncertain, they will be excluded.

Contra-indications for MRI scanning, as well as contra-indications to intra-venous administration of contrast agents were discussed with Ms. Shanta Kalaykhan-Sewradj, head of MRI technicians in the UMC Utrecht. For further information, the booklet 'Bijwerkingen van contrastmiddelen: de gadoliniumverbindingen' by Esther Ensing and Janet Hoven was used (Published by Nederlandse Vereniging voor Slachtoffers van Medische Contrastmiddelen, 2004).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients above 18 years with osteoarthritis of the knee and a future planned osteotomy of the tibia or femur are eligible for participation in this study.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
MRI T1 signal, change from baseline | Change from baseline 9 months after surgery (HTO)
  MRI T1 signal is deducted from dGEMRIC measurements

SECONDARY OUTCOMES:
KOOS clinical score, change from baseline | Change from baseline 9 months after surgery (HTO)
  Knee and Osteoarthritis Outcome Score (clinical score, completed by all participants)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Saris, MD, PhD, Study Chair — University Medical Center Utrecht, the Netherlands
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Burstein D. Tracking longitudinal changes in knee degeneration and repair. J Bone Joint Surg Am. 2009 Feb;91 Suppl 1:51-3. doi: 10.2106/JBJS.H.01412. PMID 19182025
- [Background] Brouwer RW, Bierma-Zeinstra SM, van Koeveringe AJ, Verhaar JA. Patellar height and the inclination of the tibial plateau after high tibial osteotomy. The open versus the closed-wedge technique. J Bone Joint Surg Br. 2005 Sep;87(9):1227-32. doi: 10.1302/0301-620X.87B9.15972. PMID 16129748
- [Derived] Rutgers M, Bartels LW, Tsuchida AI, Castelein RM, Dhert WJ, Vincken KL, van Heerwaarden RJ, Saris DB. dGEMRIC as a tool for measuring changes in cartilage quality following high tibial osteotomy: a feasibility study. Osteoarthritis Cartilage. 2012 Oct;20(10):1134-41. doi: 10.1016/j.joca.2012.07.001. Epub 2012 Jul 10. PMID 22796509
- See also: Affiliation site — http://www.umcutrecht.nl